CLINICAL TRIAL: NCT04122586
Title: Mechanism of PERK - eIF2a Pathways in Intestinal Mucosal Barrier of IBS-D and the Role "Metabolism Ingredients " of Tongxieyaofang
Brief Title: Mechanism of PERK - eIF2a Pathways in Intestinal Mucosal Barrier of IBS-D and the Role "Metabolism Ingredients" of Tongxieyaofang
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 81774304
Record Dates: First submitted 2019-09-25; First posted 2019-10-10 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-10

CONDITIONS: IBS (Irritable Bowel Syndrome)
Keywords: IBS-D
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- health control group (No Intervention)
- Tongxieyaofang granule group (Experimental)
  Interventions: Drug: Tongxieyaofang(granule)

INTERVENTIONS:
Drug: Tongxieyaofang(granule) — Take this granule twice a day,one bag for each time,one hour after a meal,for 4 weeks
  Arms: Tongxieyaofang granule group

SUMMARY:
Diarrhea irritable bowel syndrome(IBS-D）has seriously affected health and quality of life of patients.It may be important pathogenesis in development and recurrence of the process of IBS-D,excessive endoplasmic reticulum stress (ERS) activated PERK(proteinkinaseR-like ERkinase，PERK)-eIF2a(eukaryotic translation initiation factor 2 alpha,eIF2a) pathway and damaged intestinal mucosal epithelial Barrier. Tongxieyaofang(TXYF) had obtained satisfactory effect in treating IBS-D in clinic and previous study, but it is unknown that herbal formula how to work.This project applies metabolomics method to detect plasma,urine and stool metabolites for patients before and after treatment, to determine the effects of the"multiple ingredients"of TXYF in body.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the diagnostic criteria of Western medicine for IBS-D;
* aged 18-70 years old; with a baseline IBS-SSS score over 75 points;
* voluntarily signed the informed consent;
* local resident who could ensure follow-ups, with basic reading ability

Exclusion Criteria:

* Patients with IBS-C, -M, and uncertain forms;
* accompanied with serious lesions in major organs including heart, liver, and kidney, hematopoietic system diseases, and tumors;
* gastrointestinal organic disease (e.g., chronic pancreatitis), or systemic diseases affecting the digestive tract motion (e.g., hyperthyroidism,diabetes, chronic renal insufficiency, and nervous system diseases);
* undergoing or requiring constant use of drugs that may affect gastrointestinal functions (e.g., anti-cholinergic drugs, calcium channel blockers, 5-HT3 receptor antagonist, antidiarrheal agents, antacids, prokinetic agents, antidepressants, anxiolytics, and intestinal flora regulating drugs);
* with history of abdominal surgery (e.g., cholecystectomy);
* with an allergy history of tested drugs or severe allergy history of food;
* pregnant and lactating female;
* with a history of neurological or psychiatric disorders;
* or participating in other clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome Symptom Severity(IBS-SSS) scale | IBS-SSS was evaluated by patients at 4th week
  Patients are graded according to their own symptoms（abdominal pain，bloating，defecation satisfaction，the extent to which the disease affects the lives of patients，bowel movements）, the total score less than 75 points was considered as in remission, 75~175 as mild, 175~300 as moderate, and over 300 as severe. We will assess changes in patient scores before and after treatment to reflect the extent of disease remission.
Bristol stool form scale（BSFS） | BSFS was evaluated by patients at 4th week
  Different fecal types can reflect different intestinal transit times, the lower the score, the longer the transmission time; the higher the score, the shorter the transmission time. We will assess changes in scores before and after treatment to reflect the extent of disease remission.

SECONDARY OUTCOMES:
IBS-D PRO( patient reported outcomes) Scale | IBS-D PRO Scale was evaluated at 4th week
  Grading from the field of physiology, independence, and psychology，Use score changes to assess improvement in all areas of the patient.Minimum score is 0，means no symptoms，maximum score is 144，means all symptoms are severe.
SF-36(the MOS item short from health survey)Scale | SF-36 Scale was evaluated at 4th week
  Score evaluation from 8 aspects: physical function, role-physical, pain, global health status, vitality，social function,role-emotional， mental health.Use score changes to assess improvement in all areas of the patient. Maximum score is147.The higher the score, the better the status in all aspects.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiyuan hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided